CLINICAL TRIAL: NCT04804904
Title: A Single Center, Phase I, Open-Label, Randomized, Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of TQB3101 in Healthy Subjects
Brief Title: A Pharmacokinetic Study of TQB3101 in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TQ-B3101-I-02
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2021-03

CONDITIONS: Pharmacokinetic Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQ-B3101: Fed + Fast (Experimental): In each of the two study periods (separated by a washout period),a single dose of TQ-B3101 will be administered.Participants will receive TQ-B3101 in fed condition on Day 1 of treatment period 1 followed by a single oral dose of TQ-B3101 in fasted condition on Day 1 of treatment period 2.
  Interventions: Drug: TQ-B3101
- TQ-B3101: Fast+Fed (Experimental): In each of the two study periods (separated by a washout period),a single dose of TQ-B3101 will be administered.Participants will receive TQ-B3101 in fasted condition on Day 1 of treatment period 1 followed by a single oral dose of TQ-B3101 in fed condition on Day 1 of treatment period 2.
  Interventions: Drug: TQ-B3101

INTERVENTIONS:
Drug: TQ-B3101 — TQ-B3101 oral capsule

SUMMARY:
Evaluate the effect of food on the pharmacokinetics of TQB3101 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be willing and able to give written informed consent by signing an IRB-approved Informed Consent Form prior to admission to this study;
* Subjects must be willing and able to communicate well, understand and follow the protocol required to complete the study;
* Males and females between 18 to 60 years of age
* Males and females with a body mass Index (BMI) range 19~26 kg/m2 inclusive, male subject not less than 50kg, female subject not less than 45kg。
* Male subjects must agree to use a medically acceptable method of contraception from Screening until 6 months after administration of the last dose of study drug
* Male subjects agrees not to donate sperm for at least 6 months after administration of the last dose of study drug
* Female subjects of non-childbearing potential measures, meeting at least one of the following criteria:①menorrhoeal for 12 months and FSH >40mIU/mL;② hysterectomy;③oophorectomy.
* Subjects who are healthy as determined by physical examination,vital signs, 12-Lead ECG and X-ray examination.

Exclusion Criteria:

* Subjects who have a history or presence of cardiovascular, neurological, endocrine, respiratory, hematological, immunological, psychiatric diseases or disorders that, could affect the conduct of the study or the absorption, metabolism or excretion of the study drug.
* Subjects who have a history of relevant drug hypersensitivity or atopic allergic disease history(asthma,urticaria, eczema dermatitis).
* Current or recent (within 6 months of study drug administration) gastrointestinal , liver and kidney disease that could impact upon the absorption of study drug.
* Any major surgery within 4 weeks of study drug administration .
* Subjects who consume more than 14 units of alcohol per week during 3 months before drug administration, taken any alcohol-containing products within 24 hours ,or subjects who test negative alcohol at screening and admission
* Smokers who smoked more than 5 cigarettes before study drug administration,or can not quit smoking during the study.
* Subjects who test positive for drugs of abuse.
* Subjects who have donated blood or have a blood loss(≥300mL)within the previous 3 months prior to first dosing.
* Subjects who used any drugs that change liver enzyme activity,such as inhibitors or inducers of CYP3A4, P-gp or BCRP within 28days;
* Subjects who used any drugs including over thePrescription drugs, counter medications ,vitamin products herbal preparations.
* Subjects who have taken a special diet (including grapefruit, etc.) or exercised vigorously in the 14 days ,or other factors affecting drug absorption, distribution, metabolism, and excretion
* Participated in drug clinical trials within 3 months before taking the study ;
* Subjects with laboratory abnormalities,or or white blood cell count, neutrophil cell count and the percentage of the platelet count below the normal limit.
* Positive test result for HIV antibodies.
* Positive test for treponema Antibodies hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab).
* Subjects who have acute disease or concomitant medication at the time of screening and/or admission.
* Subjects who consuming chocolate, any caffeine-rich or xanthine-rich food or drink 24 hours before.
* The PI considered other factors unfit to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-03 (Actual)

PRIMARY OUTCOMES:
Cmax | pre-dosing on Day 1 up to 144 hours post-dosing
  maximum concentration of the analyte in plasma
Tmax | pre-dosing on Day 1 up to 144 hours post-dosing
  Time to Reach the Maximum Observed Plasma Concentration (Cmax) of the analyte
AUC0-t | pre-dosing on Day 1 up to 144 hours post-dosing
  Area Under the Concentration-time Curve From Zero (Pre-dose) to Time of Last Quantifiable Concentration of the analyte
AUC0-inf | pre-dosing on Day 1 up to 144 hours post-dosing
  Area Under the Plasma Concentration-time Curve from Time 0 to Infinite Time of the analyte

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality, China